CLINICAL TRIAL: NCT04799704
Title: Tear Film SARS-nCoV-2 Detection in Symptomatic and Pauci-symptomatic
Brief Title: Tear Film SARS-nCoV-2 Detection in Symptomatic and Pauci-symptomatic Patients.
Acronym: Eye-Covid
Status: Terminated | Type: Observational
Why Stopped: insufficient positive samples
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64002
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2022-06

CONDITIONS: Covid19; Eye Diseases
MeSH Terms: conditions — COVID-19; Eye Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- symptomatic patient: to confirm the detectability of the SARS-nCoV-2 in the tear film of symptomatic patients.
  Interventions: Diagnostic Test: swabbing of conjunctiva

INTERVENTIONS:
Diagnostic Test: swabbing of conjunctiva — Each eye will be sampled with a single, sterile, nylon, flocked swab

SUMMARY:
To investigate the presence of SARS-nCoV-2 in the tear film of symptomatic and pauci-symptomatic SARS-nCoV-2 positive patients.

DETAILED DESCRIPTION:
The end goal of the study is to show whether or not the virus can be found in the tear film in both symptomatic and less symptomatic patients by means of serial sampling.

A sample of the tears / conjunctiva will be taken with a soft brush (similar to a cotton swab) every three days until the end of the hospitalization. In addition, you must complete a questionnaire that assesses the symptoms present.

ELIGIBILITY:
Inclusion Criteria:

* Subject needs to be above 18 years old.
* The subject is willing to undergo sampling of the conjunctiva.
* The subject is willing to fill in a questionnaire.
* The subject is fluent in written and verbal Dutch.
* The subject is capable of giving informed consent.
* Applicable for part 1 only: the subject test positive for SARS-nCoV-2 on a nasopharyngeal swab. The time window between a positive nasopharyngeal swab and the first conjunctival swab may be no more than 3 days.

Exclusion Criteria:

* Allergy to Oxybuprocainehydrochloride
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: positive test for SARS-nCoV-2 on a nasopharyngeal swab.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2020-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Delbeke Heleen, MD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Result] Leysen L, Delbeke H, Desmet S, Schauwvlieghe PP, Maes P, Blanckaert G, Matthys E, Joossens M, Casteels I. In search of viable SARS-CoV-2 in the tear film: a prospective clinical study in hospitalized symptomatic patients. Clin Microbiol Infect. 2022 Aug;28(8):1172-1173. doi: 10.1016/j.cmi.2022.03.026. Epub 2022 Mar 31. No abstract available. PMID 35367365
- See also: In search of viable SARS-CoV-2 in the tear film: a prospective clinical study in hospitalized symptomatic patients. — https://doi.org/10.1016/j.cmi.2022.03.026

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conjunctival sampling will take place every three days until the day of hospital discharge.
Units Other Than Participants: swabs
Groups:
- Symptomatic Patient: The first part of our study is to confirm the detectability of the SARS-nCoV-2 in the tear film of symptomatic patients.
  swabbing of conjunctiva: Each eye will be sampled with a single, sterile, nylon, flocked swab
Period: Overall Study
Arm/Group | Symptomatic Patient
Started | 30; 176 swabs
Completed | 30; 176 swabs
Not Completed | 0; 0 swabs

BASELINE CHARACTERISTICS:
Arm/Group | Symptomatic Patient
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 30

OUTCOME MEASURES:

1. Primary Outcome: The Presence of SARS-nCoV-2 in the Tear Film of Symptomatic and Pauci-symptomatic SARS-nCoV-2 Positive Patients.
Description: Bilateral conjunctival sampling will be performed on both eyes after the application of a drop of topical anesthesia at least once.
Time Frame: during hospitalization every 3 days until the day of discharge up to 1 month
Population: symptomatic patients admitted at our University Hospital Leuven, Belgium with a positive nasopharyngeal swab for SARS-nCoV-2
Measure: Number; unit: swabs
Units Other Than Participants: swabs
Arm/Group | Symptomatic Patient
Number analyzed (Participants) | 30
Number analyzed (swabs) | 176
swabs
  positive SARS-CoV-2 swab | 13
  strongly positive SARS-CoV-2 | 3
  weakly positive SARS-CoV-2 | 10

ADVERSE EVENTS:
Time Frame: Sampling will be repeated every 3 days to evaluate if PCR becomes positive during the course of disease and to monitor the duration of detectability of the virus in tears, up to 1 month
Arm/Group | Symptomatic Patient
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT04799704/Prot_SAP_000.pdf